CLINICAL TRIAL: NCT04021394
Title: Dynamic Influence of the Epithelial-to-mesenchymal Transition (EMT) on Circulating Tumor Cell (CTC) Generation, Phenotype, and Disease Progression in Prostate Cancer
Brief Title: Influence of EMT on CTCs and Disease Progression in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Alison Allan, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: EMT Prostate
Record Dates: First submitted 2019-07-03; First posted 2019-07-16 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: circulating tumor cell; epithelial-to-mesenchymal transition; treatment response; phenotype
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-metastatic, high-risk hormone sensitive prostate cancer: Phlebotomy collection of 2 tubes of blood then annual follow up for 5 years
  Interventions: Diagnostic Test: CellSearch CTC platform; Diagnostic Test: Parsortix CTC platform
- Low-volume metastatic hormone-sensitive prostate cancer: Phlebotomy collection of 2 tubes of blood then annual follow up for 5 years
  Interventions: Diagnostic Test: CellSearch CTC platform; Diagnostic Test: Parsortix CTC platform
- High-volume metastatic hormone-sensitive prostate cancer: Phlebotomy collection of 2 tubes of blood then annual follow up for 5 years
  Interventions: Diagnostic Test: CellSearch CTC platform; Diagnostic Test: Parsortix CTC platform
- Metastatic castrate-resistant prostate cancer: Phlebotomy collection of 2 tubes of blood then annual follow up for 5 years
  Interventions: Diagnostic Test: CellSearch CTC platform; Diagnostic Test: Parsortix CTC platform

INTERVENTIONS:
Diagnostic Test: CellSearch CTC platform — epithelial-based marker approach for immunomagnetic enrichment, isolation, and quantitative immunofluorescence of CTCs
Diagnostic Test: Parsortix CTC platform — EMT-independent platform

SUMMARY:
The presence of circulating tumor cells (CTCs) in the blood of prostate cancer patients has been shown to be an important indicator of metastatic disease and poor prognosis. Additionally, changes in CTC number throughout treatment have been demonstrated to reflect therapy response. However, the CellSearch® (Menarini-Silicon Biosystems) is the only FDA- and Health Canada-cleared CTC platform available at the present time, and is thus considered the current "gold standard" for clinical CTC analysis.

Notably, CTCs are undetectable in ~35% of metastatic CRPC patients. This suggests that either CTCs are truly not present in >1/3 of patients with advanced metastatic disease; and/or that CTCs are present but not detectable as they do not meet the standard CellSearch® definition of CTCs. Given the accumulating evidence that prostate cancer cells can lose epithelial characteristics as they evolve towards a more metastatic phenotype, the investigators believe the latter scenario is most likely.

The epithelial-to-mesenchymal transition (EMT) is a critical process during embryonic development and cancer metastasis.

Although the role of androgen receptor (AR) signaling in EMT is poorly understood, studies have also demonstrated that EMT may be facilitated by androgen deprivation, castration-resistance, and/or disruption of androgen signaling.

Importantly, several clinical studies have demonstrated that CTCs with a purely mesenchymal phenotype are undetectable by CellSearch®, but that the presence of mesenchymal marker expression on CTCs with a hybrid epithelial-mesenchymal phenotype is indicative of poor prognosis. In addition, previous pre-clinical data from the Allan laboratory has demonstrated that in animal models, prostate cancers with a mesenchymal phenotype shed greater numbers of CTCs more quickly and with greater metastatic capacity than those with an epithelial phenotype. Notably, the clinically-used CellSearch®-based assay captured the majority of CTCs shed during early-stage disease in vivo, and only after the establishment of metastases were a significant number of undetectable CTCs present. This suggests that current clinical assays may be limiting ability to capitalize on the full potential of CTCs, and that a greater understanding of CTC biology is necessary in order to guide future technology development and translation to the clinic.

DETAILED DESCRIPTION:
The presence of circulating tumor cells (CTCs) in the blood of prostate cancer patients has been shown to be an important indicator of metastatic disease and poor prognosis. Additionally, changes in CTC number throughout treatment have been demonstrated to reflect therapy response. Although these cells are very rare (~1 CTC per 105-107 leukocytes), recent technological advances have now facilitated sensitive enumeration and characterization of CTCs. Techniques to enrich and analyze CTCs include size- and/or density-based separation and antibody-based techniques with/without the aid of microfluidics, while detection techniques rely almost exclusively on protein- (immunofluorescence/flow cytometry) or nucleic acid-based (RT-PCR/qRT-PCR) assays. However, the CellSearch® (Menarini-Silicon Biosystems) is the only FDA- and Health Canada-cleared CTC platform available at the present time, and is thus considered the current "gold standard" for clinical CTC analysis.

CellSearch® uses an epithelial-based marker approach for immunomagnetic enrichment, isolation, and quantitative immunofluorescence of CTCs. Using this assay, it has been demonstrated that CTCs are readily detectable in ~65% of castrate-resistant prostate cancer (CRPC) patients and that the presence of ≥5 CTCs in 7.5ml of blood is indicative of progressive metastatic disease and reduced overall survival. Notably, CTCs are undetectable in ~35% of metastatic CRPC patients. This suggests that either CTCs are truly not present in >1/3 of patients with advanced metastatic disease; and/or that CTCs are present but not detectable as they do not meet the standard CellSearch® definition of CTCs (EpCAM+/Cytokeratin 8/18/19 [CK]+/DAPI+/CD45-). Given the accumulating evidence that prostate cancer cells can lose epithelial characteristics as they evolve towards a more metastatic phenotype, the investigators believe the latter scenario is most likely.

The epithelial-to-mesenchymal transition (EMT) is a critical process during embryonic development and cancer metastasis. Activation of EMT leads to profound phenotypic changes resulting in loss of cell polarity, loss of cell-cell adhesion, resistance to apoptosis, and acquisition of migratory/invasive properties. It has also been proposed that tumor cells (via the mesenchymal-to-epithelial transition [MET]) may revert back to an epithelial phenotype in order to facilitate metastatic growth in secondary sites, suggesting a role for phenotypic plasticity during metastatic progression. At the molecular level, EMT is mediated by decreased expression of epithelial proteins (E-cadherin, CK, EpCAM); as well as corresponding increases in mesenchymal factors (N-cadherin, Vimentin, Twist, Zeb), with MET mediated by the opposite changes.

Clinically, Gleason grading can arguably be viewed as morphological evidence of EMT, since increasing Gleason score is associated with progressive loss of epithelial architecture, loss of defined basement membrane/cell polarity, and increased invasion. In support of this, studies have demonstrated that decreased expression of E-Cadherin or increased expression of mesenchymal markers (Vimentin, N-Cadherin, SNAIL) in primary prostate tumors is associated with advanced Gleason score, metastasis, and/or poor prognosis. Although the role of androgen receptor (AR) signaling in EMT is poorly understood, studies have also demonstrated that EMT may be facilitated by androgen deprivation, castration-resistance, and/or disruption of androgen signaling.

Importantly, several clinical studies have demonstrated that CTCs with a purely mesenchymal phenotype are undetectable by CellSearch®, but that the presence of mesenchymal marker expression on CTCs with a hybrid epithelial-mesenchymal phenotype is indicative of poor prognosis. In addition, previous pre-clinical data from the Allan laboratory has demonstrated that in animal models, prostate cancers with a mesenchymal phenotype shed greater numbers of CTCs more quickly and with greater metastatic capacity than those with an epithelial phenotype. Notably, the clinically-used CellSearch®-based assay captured the majority of CTCs shed during early-stage disease in vivo, and only after the establishment of metastases were a significant number of undetectable CTCs present. This suggests that current clinical assays may be limiting the ability to capitalize on the full potential of CTCs, and that a greater understanding of CTC biology is necessary in order to guide future technology development and translation to the clinic.

ELIGIBILITY:
Inclusion Criteria (all patients):

* histologically diagnosed prostate cancer
* signed informed consent

HR-HSPC cohort

* previous prostatectomy
* previous treatment with androgen deprivation therapy for <90 days and/or recommended but not yet started new line of androgen deprivation therapy
* adverse pathological findings (>=1 of extracapsular extension, positive margins, and/or seminal vesicle invasion)
* documented evidence of biochemical failure following adjuvant/salvage radiation therapy
* PSA of >1 ng/ml

LV-mHSPC cohort

* previous treatment with androgen deprivation therapy for <90 days and/or recommended but not yet started new line of androgen deprivation therapy
* documented evidence of metastatic disease (bone only; less than 4 lesions contained within the vertebral column or pelvis)

HV-mHSPC cohort

* previous treatment with androgen deprivation therapy for <90 days and/or recommended but not yet started new line of androgen deprivation therapy
* documented evidence of "high volume" metastatic disease (visceral metastases [extranodal] and/or bone metastases [>=4 bone lesions with >=1 lesion outside the vertebral column or pelvis])

mCRPC cohort

* documented evidence of progression while receiving androgen ablation therapy (medical or surgical castration) according to PCWG2 criteria
* documented evidence of metastatic disease (bone or visceral)

Exclusion Criteria:

* patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer (all cohorts)
* documented evidence of metastatic disease (HR-HSPC cohort)
* documented evidence of castrate-resistance (all HSPC cohorts)
* currently on active androgen deprivation therapy (all HSPC cohorts)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
CTC enumeration capacity | 1-2 years
  Number of CTCs as assessed by the Parsortix system versus the clinical gold standard CellSearch platform
CTC recovery capacity | 1-2 years
  Number of CTCs that can be isolated from the Parsortix system
Comparison of AR and EMT characteristics | 1-2 years
  Level of RNA expression of AR and EMT markers (EpCAM, E-Cadherin, N-Cadherin, Zeb-1) as assessed by multiplex qRT-PCR of CTCs isolated from the Parsortix system

SECONDARY OUTCOMES:
Relationship of CTC count to disease features | 1-2 years
  Differences in the number of CTCs between each of the 4 patient cohorts, and differences in the level of RNA expression of AR and EMT markers between each of the 4 patient cohorts
CTC counts and prognosis of OS and PFS | 5 years
  Correlation between number of CTCs and progression free survival and overall survival, and correlation between the level of RNA expression of AR/EMT markers and PFS and OS

CONTACTS AND LOCATIONS:
Overall Officials: Alison Allan, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No